CLINICAL TRIAL: NCT04176575
Title: Acupuncture for Pain Related to Advanced Cancer Using Dr. Tan's Balancing Method
Brief Title: Balancing Method for Pain Related to Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ronald M. Glick, MD, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY18120017
Record Dates: First submitted 2019-11-01; First posted 2019-11-25 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Pain, Cancer; Metastatic Cancer; Invasive Cancer
Keywords: Acupuncture; Cancer Pain
MeSH Terms: conditions — Cancer Pain; Neoplasm Metastasis | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This clinical trial is a descriptive, interventional, and open-label pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental): Eligible participants:
  * have advanced stage cancer and associated pain
  * will receive up to 12 acupuncture sessions
  * will attend sessions at UPMC's Center for Integrative Medicine
  * will complete study assessments at each visit
  * will complete a follow-up 4 to 6 weeks after their last acupuncture visit. Total study involvement will range from 16 to 18 weeks.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture involves inserting thin needles into precise points on the body, known as acupuncture points, for therapeutic effect. Acupuncture will be provided by a licensed acupuncturist utilizing Dr. Tan's Balancing Method.

SUMMARY:
Balancing Method for Pain Related to Advanced Cancer seeks to confirm the benefit of acupuncture for patients with pain related to advanced cancer.

DETAILED DESCRIPTION:
Pain is common among patients with cancer, with estimates as high as 90% for those with advanced disease. Opioid medication, the most common treatment, has potential adverse effects including nausea and fatigue, further interfering with quality of life. Acupuncture has been studied for the treatment of cancer-related pain, with promising results in a few methodologically sound studies with small sample size. Prior studies have found beneficial effects of open treatment using a Traditional Chinese Medicine (TCM)-based acupuncture protocol and Dr. Tan's Balancing Method. This open trial seeks to confirm the benefit of acupuncture, utilizing Dr. Tan's Balancing Method, for patients with pain related to advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Current diagnosis of a malignancy.
3. Locally invasive, metastatic, or systemic involvement from the disease, which would be anticipated to produce pain.
4. Average pain level, on a numeric rating scale, of 4/10 or higher on the Numeric Rating Scale (NRS).
5. Receiving treatment through Hillman Cancer Center, Magee Hospital, or 1 of the University of Pittsburgh Cancer Institute sites.
6. Able to read and write English.

Exclusion Criteria:

1. Experience with acupuncture within the prior 3 months.
2. Platelet count < 50,000.
3. Absolute Neutrophil Count < 1,000.
4. Treatment with anticoagulant medication, other than prophylactic levels of heparin or low molecular weight heparin preparations or anti-platelet agents.
5. Known coagulopathy.
6. Pregnancy. While it is unlikely that any patients undergoing advanced cancer treatment will be pregnant, given the lack of documented safety, this is an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Measuring effectiveness of acupuncture by assessing change in pain ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Numeric Rating Scale v.1.0 - Pain Intensity 1a (NRS) | Baseline, each visit; up to 18 weeks (per participant)
  Participant report of pain on average on a scale from 'no pain' (0) to "worst imaginable pain" (10). Higher scores mean worse outcome.
Measuring effectiveness of acupuncture by assessing change in pain intensity ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Pain Intensity Scale | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "no pain" (1) to "very severe" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing change in pain interference ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Pain Interference Short Form 4a | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "not at all" (1) to "very much" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing change in fatigue ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Fatigue Short Form 4a | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "not at all" (1) to "very much" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing change in anxiety symptom ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Emotional Distress-Anxiety - Short Form 4a | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "never" (1) to "always" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing change in sleep disturbance ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Sleep Disturbance - Short Form 4a | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "very poor/very much" (1) to "very good/not at all" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing change in gastrointestinal symptom ratings Weekly from Week 1-Week 12 and 4 week follow-up using PROMIS ® Item Bank v.1.0 measures: Gastrointestinal Nausea and Vomiting | Baseline, each week, at follow-up; up to 18 weeks (per participant)
  Participant report of symptoms in the past week on a scale from "never" (1) to "always" (5). Higher scores mean worse outcome. These measures assess changes in symptoms over the course of study participation.
Measuring effectiveness of acupuncture by assessing improvement in global symptoms ratings at Week 4 and Weeks 9-12 and 4 week follow-up using Patient Global Index of Change: Improvement (PGIC-I) | Week 5, Weeks 9-12 and follow-up; up to 18 weeks (per participant)
  Participant rating of symptom severity on a scale of -2 (much better) to 2 (much worse). Higher scores mean worse outcome. This measure assesses changes in symptoms over the course of study participation.
Measuring health intervention attitudes and beliefs at start of study by using Healing Encounters Attitudes List Measures: Treatment Expectancy (HEAL-TEX) | Baseline Visit
  Participant report of treatment expectancy on a 5 point scale (1-5) ranging from "Not at all" (1) to "Very much" (5). Higher scores ("Very much") indicate higher treatment expectancy.
Measuring perception of effectiveness based on patient-provider connections by using Healing Encounters Attitudes List: Perception of the Patient-Provider Connection (HEAL-PPC) | Week 4 and Weeks 9, 10, 11, 12
  Participant report of the patient-provider connection on a 5 point scale ranging from "Not at all" to "Very much". Higher scores ("Very much") mean better outcome. This measure assesses a change in the patient-provider connection from the beginning of study participation to the end.
Measuring spiritual attitudes and beliefs at start of study by using Healing Encounters Attitudes List Measures: Spirituality (HEAL-SPT) | Baseline Visit
  Participant report of Spirituality on a 5 point scale (1-5) ranging from "Not at all" (1) to "Very much" (5). Higher scores ("Very much") indicate higher personal spiritual belief.
Monitoring and recording use of opioids throughout the study protocol using Opioid Use Questionnaire | Baseline; weekly; follow-up; up to 18 weeks (per participant)
  Internally-developed, participant report of pain medication use. This questionnaire collects dosing/frequency information, which is used to calculate morphine equivalent dosing (MED). This information will be used to assess change in pain medication use over the course of study participation.
Assessing for treatment-related adverse events as recorded by Acupuncture Safety Record | Baseline; each visit and follow-up; up to 18 weeks (per participant)
  Internally-developed, participant report of acupuncture related adverse events. Administered in a checklist form. More selections on this form means more acupuncture related adverse events.
Assessing for treatment-related and illness-related symptoms as recorded by Symptoms Checklist (SC) | Baseline; each visit and follow-up; up to 18 weeks (per participant)
  Captures new or worsening health problems participants have experienced since their last study visit. More selections on this form means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Glick, MD, Principal Investigator — Hillman Cancer Center
Locations (1):
- UPMC Center for Integrative Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No